CLINICAL TRIAL: NCT04055714
Title: Feasibility of Balloon Dilation of the Eustachian Tubes for Dilatory Dysfunction Under Local Anesthesia
Brief Title: Feasibility of Balloon Dilation of the Eustachian Tubes Under Local Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Piedmont Ear, Nose, Throat and Related Allergy, PC (Other)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS A-016
Record Dates: First submitted 2019-08-03; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Chronic Eustachian Salpingitis
Keywords: Eustachian tube dysfunction

STUDY DESIGN:
Intervention Model Description: prospective, non-significant risk, multi-center, non-controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment arm (Experimental): Balloon dilation of the Eustachian Tube(s) with Acclarent Aera Balloon
  Interventions: Device: Balloon dilation of the Eustachian tubes

INTERVENTIONS:
Device: Balloon dilation of the Eustachian tubes — Use the Aera Balloon through the nose to dilate the Eustachian tubes

SUMMARY:
The objective of this study is to demonstrate that balloon dilation of the Eustachian tubes can be done successfully for treatment of chronic dilatory Eustachian tube dysfunction under local anesthesia with acceptable patient discomfort levels.

DETAILED DESCRIPTION:
This study is a prospective, non-significant risk, multi-center trial of patients with Eustachian tube dysfunction who are refractory to medical management. Patients will undergo balloon dilation of the Eustachian tubes in the office under local anesthesia. We will assess assess the peri-procedural and post-procedure pain levels, and determine the proportion of subjects experiencing normalization of tympanometry and improvement in quality of of life at 6 weeks, 12 weeks, and 52 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female aged 22 years and older
2. Persistent ETD as defined by patient-reported symptoms of ETD (including pressure and/or pain and/or clogged and/or muffled sensation in the affected ear(s)) for no less than 12 weeks prior to enrollment, and at least one of the following confirmatory indicators of persistent ETD no less than 12 weeks prior to enrollment B1: Confirmation from referring physician that the subject has experienced persistent ETD symptoms (including pressure and/or pain and/or clogged and or muffled sensation in the affected ear(s)) during an office visit no less than 12 weeks prior to enrollment. Persistent symptoms must be confirmed as not waxing and waning. OR B2: Documented evidence in the ENT physician records that the subject has experienced persistent ETD symptoms (including pressure and/or pain and/or clogged and/or muffled sensation in the affected ear(s)) during an office visit no less than 12 weeks prior to enrollment. Persistent symptoms must be confirmed as not waxing and waning. OR B3: Type B or Type C tympanogram in at least one ear no less than 12 weeks prior to enrollment. OR B4: Otoscopic exam demonstrating TM retraction and/or middle ear fluid no less than 12 weeks prior to enrollment.
3. Failure of appropriate medical management consisting of either a minimum of 4 weeks of continuous daily usage of any intranasal steroid spray (INS) or a minimum of one completed course of an oral steroid, per the investigator's choice. The failed medical management may occur any time within 90 days prior to study enrollment.
4. A positive diagnosis of persistent (i.e. not waxing and waning) ETD, as confirmed with both of the following:

   D1: Abnormal tympanometry (defined as either Type B or Type C) after failed medical management and within 14 days of study enrollment D2: Symptomatic dysfunction as documented by a Eustachian Tube Dysfunction Questionnaire (ETDQ-7) mean item score ≥ 2.1 after failed medical management
5. Absence of internal carotid artery (ICA) dehiscence into the ET lumen on both sides as confirmed by a computed tomography (CT scan) including temporal bone - to include paranasal sinuses when clinically appropriate

Exclusion Criteria:

1. Females who are pregnant or lactating
2. Anatomy that requires an adjunctive surgical procedure on the same day as ETBC surgery to allow balloon catheter access to the ET (e.g. septoplasty, polypectomy, turbinate reduction)
3. Concomitant nasal or sinus procedures planned on the same day as ETBC surgery or any time during study participation (e.g. adenoidectomy, sinus surgery)
4. Concomitant ear procedures planned on the same day as ETBC surgery or any time during study participation (e.g. myringotomy, tympanostomy tube placement)
5. History of major surgery of the head or neck within four (4) months prior to enrollment (e.g. adenoidectomy, sinus surgery)
6. History of a patulous ET in either ear
7. History of fluctuating sensorineural hearing loss, in either ear, within the past 5 years, as evidenced by a 20dB change in 3 pure tone average frequencies
8. Active chronic or acute otitis media (AOM), in either ear, as evidenced by bulging TM, erythema, purulent effusion, or cholesteatoma
9. Tympanic membrane perforation or presence of a tympanostomy tube in either ear
10. Tympanosclerosis with opacification of ≥50% of tympanic membrane in either ear
11. Evidence of acute upper respiratory infection
12. Evidence of active Temporomandibular joint disorder (TMJ) per clinical exam (i.e. pain with mouth opening, chewing, clenching; tenderness to palpation deep into the glenoid capsule on wide mouth opening, especially with right and left lateral movements of the jaw; tenderness of the masseter or lateral pterygoid muscles on bimanual intra/extraoral examination)
13. Cleft palate or history of cleft palate repair
14. Craniofacial syndrome, including Down's Syndrome
15. Cystic fibrosis
16. Ciliary dysmotility syndrome
17. Other systemic mucosal diseases or immunodeficiency disorders (e.g. Samters triad, Sarcoidosis, Wegener's granulomatosis), including patients actively taking immunosuppressive drugs
18. Intolerance of protocol-defined medication regimen
19. Prior surgical intervention on Eustachian tube including balloon dilation, laser or mechanical tuboplasty
20. Absence of dilatory muscular contractions (tensor veli palatini or levator veli palatini failure, severe dysfunction) as assessed by endoscopic observation of swallows and yawns
21. Treatment is planned for one ear, but the opposite ear has normal (Type A) tympanogram and the subject complains of ETD symptoms in that ear
22. Treatment is planned for one ear, but the opposite ear has abnormal (Type B or C) tympanogram and the subject has no complaints of ETD symptoms in that ear (asymptomatic)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Visual Pain Assessment Scale to describe procedural pain | during procedure
  Assess peri-procedural pain levels with a visual pain assessment scale. The scale has numbering from 0-10 with associated visual pictures that correspond to the degree of pain. Participants will number their pain level and describe the location of pain (ear, nose, forehead, jaw, teeth).
Visual Pain Assessment Scale to describe postoperative pain | 2 weeks after procedure
  Assess post-procedural pain levels with a visual pain assessment scale. The scale has numbering from 0-10 with associated visual pictures that correspond to the degree of pain. Participants will number their pain level and describe the location of pain (ear, nose, forehead, jaw, teeth).
Visual Pain Assessment Scale to describe postoperative pain | 6 weeks after procedure
  Assess post-procedural pain levels with a visual pain assessment scale. The scale has numbering from 0-10 with associated visual pictures that correspond to the degree of pain. Participants will number their pain level and describe the location of pain (ear, nose, forehead, jaw, teeth).
Visual Pain Assessment Scale to describe postoperative pain | 52 weeks after procedure
  Assess post-procedural pain levels with a visual pain assessment scale. The scale has numbering from 0-10 with associated visual pictures that correspond to the degree of pain. Participants will number their pain level and describe the location of pain (ear, nose, forehead, jaw, teeth).

SECONDARY OUTCOMES:
Tympanometry - an objective measure of the negative pressure in the middle ear | 6 weeks after procedure
  proportion of subjects experiencing normalization of tympanometry post-treatment, indicating improvement or resolution in the negative pressure in the middle ear.
Tympanometry - an objective measure of the negative pressure in the middle ear | 52 weeks after procedure
  proportion of subjects experiencing normalization of tympanometry post-treatment, indicating improvement or resolution in the negative pressure in the middle ear.

OTHER OUTCOMES:
Quality of life assessment using the ETDQ-7 questionnaire | 6 weeks after procedure
  Determine the proportion of subjects achieving improvement of 0.5 points at 6 weeks post-treatment, indicating significant improvement in the quality of life with respect to symptoms of Eustachian tube dysfunction.
Quality of life assessment using the ETDQ-7 questionnaire | 52 weeks after procedure
  Determine the proportion of subjects achieving improvement of 0.5 points at 6 weeks post-treatment, indicating significant improvement in the quality of life with respect to symptoms of Eustachian tube dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hoffmann, MD, Principal Investigator — Piedmont Ear, Nose, Throat & Related Allergy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swords C, Smith ME, Patel A, Norman G, Llewellyn A, Tysome JR. Balloon dilatation of the Eustachian tube for obstructive Eustachian tube dysfunction in adults. Cochrane Database Syst Rev. 2025 Feb 26;2(2):CD013429. doi: 10.1002/14651858.CD013429.pub2. PMID 40008607